CLINICAL TRIAL: NCT05790473
Title: Artificial Intelligence Algorithm for the Screening of Abnormal Fetal Brain Findings at First Trimester Ultrasound Scan
Acronym: AIRFRAME
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Ministero della Salute, Italy (Other); Azienda Ospedaliero-Universitaria di Parma (Other); Ospedale Di Venere, ASL BA, Bari Italy (Unknown)
Responsible Party: Principal Investigator, Familiari Alessandra, Clinician, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5526
Record Dates: First submitted 2023-03-06; First posted 2023-03-30 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Fetal Anomaly; Brain Malformation
MeSH Terms: conditions — Congenital Abnormalities | interventions — Artificial Intelligence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Fetuses with brain anomalies
  Interventions: Diagnostic Test: Artificial Intelligence
- Controls: Normal with normal brain
  Interventions: Diagnostic Test: Artificial Intelligence

INTERVENTIONS:
Diagnostic Test: Artificial Intelligence — Development of AI algorithm for early detection of fetal brain anomalies in the first trimester of pregnancy

SUMMARY:
Visualization of the posterior fossa brain spaces, their spatial relationship and measurements can be obtained in the midsagittal view of fetal head, the same used for NT measurement (9), and plays an important role in the early diagnosis of neural tube defects, such as open spinal dysraphism (5), and posterior fossa anomalies, such as DWM or BPC (7). However, assessment of the fetal posterior fossa in the first trimester is still challenging due to several limitations including involuntary movements of the fetus and small size of the brain structures, causing difficulties for examination and misdiagnosis. Moreover, it is also operator-dependent for the acquirement of high-quality ultrasound images, standard measurements, and precise diagnosis.

The use of new technologies to improve the acquisition of images, to help automatically perform measurements, or aid in the diagnosis of fetal abnormalities, may be of great importance for the optimal assessment of the fetal brain, particularly in the first trimester (10). Artificial intelligence (AI) is described as the ability of a computer program to perform processes associated with human intelligence, such as learning, thinking and problem-solving. Deep Learning (DL), a subset of Machine Learning (ML), is a branch of AI, deﬁned by the ability to learn features automatically from data without human intervention. In DL, the input and output are connected by multiple layers loosely modeled on the neural pathways of the human brain. In the image recognition field, one of the most promising type of DL networks is represented by convolutional neural networks (CNN). These are designed to extract highly representative image features in a fully automated way, which makes them applicable to diagnostic decision-making.

According to these observations, we propose a research project aimed to develop an ultrasound-based AI-algorithm, which is capable to assess the fetal posterior fossa structures during the first trimester ultrasound scan and discriminate between normal and abnormal findings through a fully automatic data processing.

DETAILED DESCRIPTION:
The application of AI in obstetric ultrasound includes three aspects: structure identification, automatic and standardized measurements, and classification diagnosis. Since obstetric ultrasound is time-consuming, the use of AI could also reduce examination time and improve workflow.

Study design: this is a multicenter retrospective observational cohort study and subsequent prospective cohort study. The study design will be organized in two different phases.

The first phase, the feasibility retrospective study, has the objective to develop and train AI-Algorithm with normal and abnormal images retrospectively acquired during first trimester ultrasound scan from ten international fetal medicine centers.

The second phase, a prospective clinical validation, has the objective to test the AI-Algorithm in the assessment of the fetal posterior fossa anatomy in a real clinic setting with real patients from each of the participating fetal medicine centers.

Setting: Three (3) fetal medicine centers.

Participants: singleton pregnant population who underwent ultrasound examination between 11 - 14 weeks of gestation in ten fetal medicine centers.

Primary endpoint: To validate a novel AI-based technology, which could potentially be used as a screening tool for fetal brain abnormal findings in the first trimester.

Secondary endpoints: To improve the performance of the standard first trimester screening of fetal posterior fossa ensuring its reliable sonographic assessment within a shorter time of execution. To detect higher repeatability and reproducibility, allowing to implement the ultrasound screening also in terms of efficiency on a vast scale, optimizing healthcare resources In the first phase of the study, participating fetal medicine centers will search their electronic databases for midsagittal images of singleton pregnant women who underwent ultrasound imaging at 11+0 - 13+6 weeks of gestation with any fetal posterior fossa anomaly, such as open spinal dysraphism, DWM or BPC. Normal images of the fetal posterior fossa at the same gestational age will be provided by the promoting centers - i.e., Fondazione Policlinico A. Gemelli, IRCCS and University of Parma. Clinical, ultrasound, prenatal and postnatal information of each case will be retrieved from patient's medical records and entered an electronic database collection file by the principal investigator from each participating center. The acquired images will be anonymized, saved as DICOM and shared through a dedicated cloud storage system which will be set up by the bioengineering team. Each center will be able to access the web system using a personal ID and password.

In the second phase of the study, the algorithm will be prospectively tested and validated in a real clinical setting with real patients from each of the participating fetal medicine centers. Inclusion and exclusion criteria, imaging protocol and data collection will be the same carried out during the retrospective phase.

ELIGIBILITY:
Inclusion Criteria:

* Women with single pregnancies who underwent ultrasound examination between 11+0 - 13+6 weeks of gestation or a fetal crown-rump-length between 45 - 84 mm.

Exclusion Criteria:

* Women who did not have the first trimester screening scan at the settled gestational age.
* Women in which a good visualization of the mid-sagittal view of the fetal head was not technically possible.
* Women who are not able to give the informed consent.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Study Population: All pregnancies undergoing first trimester screening
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
AI algorithm | 2 years
  Number of cases detected with AI algorithm application

SECONDARY OUTCOMES:
Reproducibility | 1 year
  Number of cases detected with AI algorithm application compared with those detected with standard techniques of prenatal diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Familiari, MD, Principal Investigator — Fondazione Policlinico Agostino Gemelli
Locations (1):
- FP Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
DICOM images through a drive among the centres
Supporting Information: Study Protocol, SAP
Time Frame: after 1 year and for 1 year
Access Criteria: pathological cases

REFERENCES:
- [Background] Garcia-Rodriguez R, Garcia-Delgado R, Romero-Requejo A, Medina-Castellano M, Garcia-Hernandez JA, Gonzalez-Martin JM, Sepulveda W. First-trimester cystic posterior fossa: reference ranges, associated findings, and pregnancy outcomes. J Matern Fetal Neonatal Med. 2021 Mar;34(6):933-942. doi: 10.1080/14767058.2019.1622673. Epub 2019 Jun 4. PMID 31113257
- [Background] Chaoui R, Benoit B, Mitkowska-Wozniak H, Heling KS, Nicolaides KH. Assessment of intracranial translucency (IT) in the detection of spina bifida at the 11-13-week scan. Ultrasound Obstet Gynecol. 2009 Sep;34(3):249-52. doi: 10.1002/uog.7329. PMID 19705402
- [Background] Drukker L, Noble JA, Papageorghiou AT. Introduction to artificial intelligence in ultrasound imaging in obstetrics and gynecology. Ultrasound Obstet Gynecol. 2020 Oct;56(4):498-505. doi: 10.1002/uog.22122. PMID 32530098
- [Background] Chen Z, Liu Z, Du M, Wang Z. Artificial Intelligence in Obstetric Ultrasound: An Update and Future Applications. Front Med (Lausanne). 2021 Aug 27;8:733468. doi: 10.3389/fmed.2021.733468. eCollection 2021. PMID 34513890

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT05790473/Prot_SAP_000.pdf